CLINICAL TRIAL: NCT01446926
Title: Safety and Immunogenicity of Pneumococcal Protein Vaccine (PPrV) in Healthy Adults, Toddlers and Infants in Bangladesh
Brief Title: Study of Investigational Pneumococcal Vaccine in Healthy Adults, Toddlers and Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PPR02; U1111-1117-7316 (Other: WHO)
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Pneumonia; Pneumococcal Infections; Streptococcus Pneumoniae Infections
Keywords: Pneumonia; Pneumococcal Infections; Streptococcus pneumoniae Infections; Pneumococcal vaccines
MeSH Terms: conditions — Pneumonia; Pneumococcal Infections | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (11):
- Group 1: Adults High Dose (Formulation 1) (Experimental): Adults who will receive a single injection of high dose investigational Pneumococcal vaccine
  Interventions: Biological: Pneumococcal Vaccine High Dose (Formulation 1)
- Group 2: Adults Placebo (Placebo Comparator): Adult participants who will receive an injection of placebo
  Interventions: Biological: Tris buffered saline (Placebo)
- Group 3: Toddlers High Dose (Formulation 1) (Experimental): Toddlers who will receive a single injection of high dose Pneumococcal vaccine
  Interventions: Biological: Pneumococcal Vaccine High Dose (Formulation 1)
- Group 4: Toddlers Placebo (Placebo Comparator): Toddlers who will receive a single injection of placebo
  Interventions: Biological: Tris buffered saline (Placebo)
- Group 5: Infants Low Dose (Formulation 2) (Experimental): Infants who will receive 3 injections of low dose low dose Pneumococcal vaccine
  Interventions: Biological: Pneumococcal Vaccine Low Dose (Formulation 2)
- Group 6: Infants Placebo (Placebo Comparator): Infants who will receive 3 injections of placebo
  Interventions: Biological: Tris buffered saline (Placebo)
- Group 7: Infants Middle Dose (Formulation 3) (Experimental): Infants who will receive 3 injections of middle dose Pneumococcal vaccine
  Interventions: Biological: Pneumococcal Vaccine Middle Dose (Formulation 3)
- Group 8: Infants Middle Dose (Formulation 4) (Experimental): Infants who will receive 3 injections of middle dose Pneumococcal vaccine
  Interventions: Biological: Pneumococcal Vaccine Middle Dose (Formulation 4)
- Group 9: Infants Placebo (Placebo Comparator): Infants who will receive 3 injections of placebo
  Interventions: Biological: Tris buffered saline (Placebo)
- Group 10: Infants High Dose (Formulation 1) (Experimental): Infants who will receive 3 injections of high dose Pneumococcal vaccine
  Interventions: Biological: Pneumococcal Vaccine High Dose (Formulation 1)
- Group 11: Infants Placebo (Placebo Comparator): Infants who will receive 3 injections of placebo
  Interventions: Biological: Tris buffered saline (Placebo)

INTERVENTIONS:
Biological: Pneumococcal Vaccine High Dose (Formulation 1) — 0.5 mL, Intramuscular
  Arms: Group 1: Adults High Dose (Formulation 1)
Biological: Tris buffered saline (Placebo) — 0.5 mL, Intramuscular
  Other Names: Tris buffered saline
  Arms: Group 2: Adults Placebo
Biological: Pneumococcal Vaccine High Dose (Formulation 1) — 0.5 mL, Intramuscular
  Arms: Group 3: Toddlers High Dose (Formulation 1)
Biological: Tris buffered saline (Placebo) — 0.5 mL, Intramuscular
  Other Names: Tris buffered saline
  Arms: Group 4: Toddlers Placebo
Biological: Pneumococcal Vaccine Low Dose (Formulation 2) — 0.5 mL, Intramuscular
  Arms: Group 5: Infants Low Dose (Formulation 2)
Biological: Tris buffered saline (Placebo) — 0.5 mL, Intramuscular
  Other Names: Tris buffered saline
  Arms: Group 6: Infants Placebo
Biological: Pneumococcal Vaccine Middle Dose (Formulation 3) — 0.5 mL, Intramuscular
  Arms: Group 7: Infants Middle Dose (Formulation 3)
Biological: Pneumococcal Vaccine Middle Dose (Formulation 4) — 0.5 mL, Intramuscular
  Arms: Group 8: Infants Middle Dose (Formulation 4)
Biological: Tris buffered saline (Placebo) — 0.5 mL, Intramuscular
  Other Names: Tris buffered saline
  Arms: Group 9: Infants Placebo
Biological: Pneumococcal Vaccine High Dose (Formulation 1) — 0.5 mL, Intramuscular
  Arms: Group 10: Infants High Dose (Formulation 1)
Biological: Tris buffered saline (Placebo) — 0.5 mL, Intramuscular
  Other Names: Tris buffered saline
  Arms: Group 11: Infants Placebo

SUMMARY:
This study is designed to explore the safety and tolerability of an investigational pneumococcal vaccine through a step-down enrollment.

Primary Objective:

* To evaluate the safety and tolerability of an investigational pneumococcal vaccine.

Secondary Objective:

* To evaluate the immunogenicity of an investigational pneumococcal vaccine.

DETAILED DESCRIPTION:
All adult participants will receive a single injection of study vaccine or placebo. After satisfactory safety evaluation, toddler participants will receive a single injection of study vaccine or placebo. After satisfactory safety evaluation, infant participants will receive 3 injections of study vaccine or placebo in dose-ascending order (low, medium, and high dose), with a safety evaluation after each dose level before the study proceeds to the next higher dose. All participants will undergo immunogenicity testing and monitoring for safety.

ELIGIBILITY:
Inclusion Criteria:

Adults:

* Aged 18 to 50 years on the day of inclusion.
* Informed consent form has been signed and dated. If the subject is unable to read the informed consent form, a site-defined standard procedure will be followed to ensure subject understanding of the process and will be marked by the subject and signed by a witness.
* Able to attend all scheduled visits and to comply with all trial procedures.

Infants and Toddlers:

* Aged 6 to 7 weeks (42 to 49 days) for infants and 12 to 13 months for toddlers on the day of inclusion
* Born at full term of pregnancy (≥37 weeks) and having a weight ≥ 60% of the median weight for Bangladesh as measured by the "weight-to-length" index.
* Informed consent form has been signed and dated by the parent(s) or other legally acceptable representative (and by an independent witness if required by local regulations). If the subject's parent(s) or other legally acceptable representative is unable to read the informed consent form, a procedure will be followed to ensure his/her understanding of the process and will be marked by the subject's parent(s) or other legally acceptable representative and signed by a witness.
* Subject and parent/guardian are able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* (Adults only): Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination).
* Participation or planned participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial vaccination except if non-interventional follow-up for an earlier study (e.g., long-term surveillance).
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination, or planned receipt of any vaccine in the 4 weeks following the trial vaccination.
* Previous vaccination against S. pneumoniae (in the previous 5 years).
* History of pneumococcal infection (confirmed microbiologically) within 5 years.
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances.
* Bleeding disorder, including thrombocytopenia contraindicating intramuscular (IM) vaccination, or receipt of anticoagulants in the 3 weeks preceding inclusion.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* (Adults only): Identified as employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the employees or the Investigator.
* (Infants and Toddlers only): Parents or guardians identified as employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the employees or the Investigator.
* Febrile illness (temperature ≥38.0°C) or moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination.
* Receipt of oral or injected antibiotic therapy within 72 hours prior to any blood draw (for immunogenicity assessment).

Ages: 6 Weeks to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 280 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants reporting solicited injection site and systemic reactions, unsolicited systemic reactions, and serious adverse events following vaccination. | Day 0 through Day 90 post-vaccination
  Solicited injection site reactions: For adults: Pain, Erythema, and Swelling; Toddlers and infants: Tenderness, Erythema, Swelling. Solicited systemic reactions: For adults, Fever (Temperature), Headache, Malaise, and Myalgia; Toddlers and infants, Fever (Temperature), Vomiting, Crying Abnormal, Drowsiness, Appetite Loss, Irritability.

SECONDARY OUTCOMES:
Immunogenicity of the Pneumococcal Vaccine in adults and toddlers | Day 30 post-vaccination (adults and toddlers)
  Evaluation of immune responses to antigen component of the investigational vaccine by enzyme-linked immunosorbent assay (ELISA).
Immunogenicity of the Pneumococcal Vaccine in toddlers | Day 30 post-vaccination 2 and 3 (infants)
  Evaluation of immune responses to antigen component of the investigational vaccine by enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Dhaka, Bangladesh

REFERENCES:
- [Result] Brooks WA, Chang LJ, Sheng X, Hopfer R; PPR02 Study Team. Safety and immunogenicity of a trivalent recombinant PcpA, PhtD, and PlyD1 pneumococcal protein vaccine in adults, toddlers, and infants: A phase I randomized controlled study. Vaccine. 2015 Aug 26;33(36):4610-7. doi: 10.1016/j.vaccine.2015.06.078. Epub 2015 Jul 2. PMID 26143615